CLINICAL TRIAL: NCT05887336
Title: Intra-Nasal Mechanical Stimulation (INMEST) As a Treatment Method for the Relief of Symptoms of Dry Eye - a Prospective, Double-blind, Pivotal Study to Evaluate the Safety and Performance of the Walther System
Brief Title: Intra-Nasal Mechanical Stimulation (INMEST) As a Treatment Method for the Relief of Symptoms of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abilion Medical Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-DE-002
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Pivotal, double-blind, randomized, multicentre study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational device treament and standard treatment (Active Comparator): After an initial demonstration of the device, study subjects will be given the device to be used for self-administration at home, 10 minutes per day in each nasal cavity, 3 days a week, for a total treatment period of six weeks.
  Interventions: Device: Walther System; Drug: Non preserved ocular lubricants; Procedure: Eye lid procedure
- Sham device treatment and standard treatment (Sham Comparator): After an initial demonstration of the device, study subjects will be given the device to be used for self-administration at home, 10 minutes per day in each nasal cavity, 3 days a week, for a total treatment period of six weeks.
  Interventions: Device: Sham Walther System; Drug: Non preserved ocular lubricants; Procedure: Eye lid procedure

INTERVENTIONS:
Device: Walther System — Walther System providing INMEST treatment
  Arms: Investigational device treament and standard treatment
Device: Sham Walther System — Walther System not providing INMEST treatment, but otherwise behave as the active comparator.
  Arms: Sham device treatment and standard treatment
Drug: Non preserved ocular lubricants — * Hyaluronic acid (HyloGel)
  * Hyaluronic acid and Ectoin (Hylo Dual Intense)
  * Hyaluronic acid and Trehalos (Theloz Duo)
Procedure: Eye lid procedure — Lid hygiene, warm eye bag, lid massage and Omega 3

SUMMARY:
The purpose of the study is to investigate the degree of symptom relief in people with signs or symptoms of dry eyes after self-treatment at home with the Walther System delivering INMEST (intranasal mechanical stimulation).

A total of 110 subjects are planned to be enrolled and randomized to either use an active device or a sham device. Both groups will also receive standard treatment in mainstream healthcare for symptoms of dry eye. The subject self-administer treatments at home, three times a week for six weeks, with a follow-up period of three months after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. The study subject reports having understood and signed the Informed Consent Form (ICF) and is willing to comply with all investigation visits and assessments
3. History of dry eye in both or one eye, supported by a previous clinical diagnosis or have self-reported history of complaints for at least 4 months prior to enrolment
4. Women of childbearing potential must agree to use a reliable, medically approved form of contraception during the study participation until end of study
5. OSDI score > 15
6. Non-Invasive tear Break-Up Time (NIBUT) ≤ 10 seconds
7. Anticipated compliance with prescribed treatment and follow-up

Exclusion Criteria:

1. Recently (3 months prior enrolment) undergone nasal or sinus surgery
2. Women who are pregnant as determined by urine test at inclusion and prior to study start (applies to sites in Denmark only)
3. Ongoing acute upper respiratory tract infection, per the Investigator's judgement
4. Bleph-ex treated within 3 months prior to enrolment
5. The study subject has a cognitive incapacity or language barrier precluding adequate understanding or cooperation
6. The study subject is considered by the Investigator to be unsuitable to participate in the investigation for any other reason
7. Any severe diseases interfering with the performance, evaluation, and outcome of the clinical evaluation
8. Previous (within 30 days prior to enrolment/randomization) and concurrent treatment during the treatment phase with another investigational drug/s or device/s

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) | Treatment period, up to 6 weeks
  Change in Ocular Surface Disease Index (OSDI) evaluated at baseline and end of treatment.

SECONDARY OUTCOMES:
Adverse Events | Study period, up to 4.5 months
  Number of treatment related Adverse Events/Adverse Device Effects/Serious Adverse Events/Serious Adverse Device Effects and Unanticipated Serious Adverse Device Effects when using the Walther System.
Device Deficiencies | Treatment period, up to 6 weeks
  Number of Walther System Device Deficiencies.
Remission | Treatment period, up to 6 weeks
  Remission of estimated symptoms with OSDI after a treatment period of 6 weeks evaluated as a binary endpoint.
Non-Invasive Tear Break-Up time (NIBUT) | Treatment period, up to 6 weeks
  Degree of increased Non-Invasive tear Break-Up time. Baseline result compared to result measured during treatment period.
Schirmer's Test | Treatment period, up to 6 weeks
  Degree of improvement of tear production according to Schirmer's test. Baseline result compared to result measured during treatment period.
Tear Meniscus Height (TMH) | Treatment period, up to 6 weeks
  Degree of change in TMH value. Baseline value compared to value measured during treatment period.
Lissamine Green Test | Treatment period, up to 6 weeks
  Lissamine green test scale changes. Baseline scale compared with scale measured during treatment period.
Corneal Staining Test | Treatment period, up to 6 weeks
  Corneal Staining test scale changes. Baseline scale compared with scale measured during treatment period.
Lipid Layer Test | Treatment period, up to 6 weeks
  Degree of improvement of Lipid Layer coverage and thickness. Baseline result compared to results measured during the treatment period.
  The test is performed with a specific interference camera that visualizes the pre corneal lipid layer spread. The Interference colour chart allows quantification of the interference images, which are graded corresponding to lipid layer thickness and coverage. Images are classified from 5 grades; 1. Open meshwork, 2. Open to closed meshwork, 3. Closed to open meshwork, 4 Closed meshwork, 5. Colour fringe
Non-Invasive Tear Break-Up time (NIBUT) | Follow-up period, up to 1 month
  Degree of increased Non-Invasive tear Break-Up time evaluated at 1 month after end of treatment period.
Non-Invasive Tear Break-Up time (NIBUT) | Follow-up period, up to 3 months
  Degree of increased Non-Invasive tear Break-Up time evaluated at 3 months after end of treatment period.
Schirmer's Test | Follow-up period, up to 1 month
  Degree of improvement of tear production according to Schirmer's test evaluated at 1 month after end of treatment period.
Schirmer's Test | Follow-up period, up to 3 months
  Degree of improvement of tear production according to Schirmer's test evaluated at 3 months after end of treatment period.
Tear Meniscus Height (TMH) | Follow-up period, up to 1 month
  Degree of change in TMH value evaluated at 1 month after end of treatment period.
Tear Meniscus Height (TMH) | Follow-up period, up to 3 months
  Degree of change in TMH value evaluated at 3 months after end of treatment period.
Lissamine Green Test | Follow-up period, up to 1 month
  Lissamine green test scale changes evaluated at 1 month after end of treatment period.
Lissamine Green Test | Follow-up period, up to 3 months
  Lissamine green test scale changes evaluated at 3 months after end of treatment period.
Corneal Staining Test | Follow-up period, up to 1 month
  Corneal Staining test scale changes evaluated at 1 month after end of treatment period.
Corneal Staining Test | Follow-up period, up to 3 months
  Corneal Staining test scale changes evaluated at 3 months after end of treatment period.
Lipid Layer Test | Follow-up period, up to 1 month
  Degree of improvement of Lipid Layer coverage and thickness evaluated at 1 month after end of treatment.
  The test is performed with a specific interference camera that visualizes the pre corneal lipid layer spread. The Interference colour chart allows quantification of the interference images, which are graded corresponding to lipid layer thickness and coverage. Images are classified from 5 grades; 1. Open meshwork, 2. Open to closed meshwork, 3. Closed to open meshwork, 4 Closed meshwork, 5. Colour fringe
Lipid Layer Test | Follow-up period, up to 3 months
  Degree of improvement of Lipid Layer coverage and thickness evaluated at 3 months after end of treatment.
  The test is performed with a specific interference camera that visualizes the pre corneal lipid layer spread. The Interference colour chart allows quantification of the interference images, which are graded corresponding to lipid layer thickness and coverage. Images are classified from 5 grades; 1. Open meshwork, 2. Open to closed meshwork, 3. Closed to open meshwork, 4 Closed meshwork, 5. Colour fringe
Compliance | Study period, up to 4.5 months
  Grade of compliance/adherence to prescribed treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Källmark, PhD, Principal Investigator — Källmarkskliniken
Locations (3):
- Denmark (2):
  - Øjenhospitalet Danmark, Charlottenlund, Copenhagen
  - Kontaktlinse Instituttet, Aarhus, Århus
- Källmarkskliniken, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No